CLINICAL TRIAL: NCT02509533
Title: Comparison of the Use of VAC (Vacuum Assisted Closure) System in Transplants of Leg Ulcers Versus Usual Dressing Method. A Monocentric, Prospective, Randomized, Parallel Groups Study
Brief Title: Comparison of the Use of VAC System in Transplants of Leg Ulcers Versus Usual Dressing Method
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties to recruit patients.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1008042; 2010-A00371-38 (Other: ANSM)
Record Dates: First submitted 2015-07-21; First posted 2015-07-28 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Leg Ulcer
Keywords: Vacuum Assisted Closure
MeSH Terms: conditions — Leg Ulcer | interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- V.A.C.® Therapy (Experimental): In this arm, investigators will use the V.A.C.® Therapy after a transplants of leg ulcers.
  Interventions: Device: V.A.C.®
- usual dressing method (compresses) (Active Comparator): In this arm, investigators will use the usual dressing method after a transplants of leg ulcers.
  Interventions: Device: dressing

INTERVENTIONS:
Device: V.A.C.® — Patients received V.A.C.® Therapy (KCI medical) after a transplants of leg ulcers.
  Arms: V.A.C.® Therapy
Device: dressing — Patients received usual dressing method (compresses) after a transplants of leg ulcers
  Arms: usual dressing method (compresses)

SUMMARY:
To evaluate the VAC (Vacuum Assisted Closure) therapy in transplants of leg ulcers versus usual dressing method. The VAC Therapy system consists of:

* A unit delivering a precise under atmospheric pressure, controlled and regulated in the wound site,
* Consumables necessary for the implementation of the dressing,
* Collecting tanks exudates with gel. VAC therapy is a system using negative pressure. It is known to be efficient into care of chronic wounds and ulcerous wounds by increasing the cicatrisation.

This system is systematically used into the dermatology unit of the CHU of Saint-Etienne after transplants of leg ulcers, but no data confirms the interest of this method compared to usual dressing method. This study will provide this data.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized into the dermatology unit
* patient with an evolutive leg ulcer since more than 1 month
* signed informed consent

Exclusion Criteria:

* known allergy to one of dressings used in this study
* patient with a non-treated osteomyelitis
* patient with tumoral tissues into the wound
* patient with raw organ or raw blood vessels
* patient with an anticoagulation treatment with a potentially hemorrhagic curative dose
* patient having hemostasis problems that can lead to hemorrhagic exudates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Percentage of healing between VAC system and compresses for all types of leg ulcers | 1 month after the transplant
  Number of patients having a wound at least 50% of the grafted area between VAC system and compresses

SECONDARY OUTCOMES:
Percentage of healing between VAC system and compresses for all types of leg ulcers | 3 months after the transplant
  Number of patients having a wound at least 50% of the grafted area between VAC system and compresses
Evolution of the pain by Analogic Visual Scale. | day 0 : just before the transplant
  Pain score as measured by visual analog scale between VAC system and compresses
Evolution of the pain by Analogic Visual Scale. | day 1 : the day after the transplant
  Pain score as measured by visual analog scale between VAC system and compresses
Evolution of the pain by Analogic Visual Scale | Month 1
  Pain score as measured by visual analog scale between VAC system and compresses
Quality of life questionnaire score. | day 0 : just before the transplant
  Quality of life questionnaire score between VAC system and compresses
Quality of life questionnaire score. | Day 5
  Quality of life questionnaire score between VAC system and compresses
Quality of life questionnaire score. | Month 1
  Quality of life questionnaire score between VAC system and compresses
Quality of life questionnaire score. | Month 3
  Quality of life questionnaire score between VAC system and compresses
Cost of the treatment. | Month 3
  Cost of the treatment, between VAC system and compresses This coast includes costs of consumables, hospitalisation days and nursing costs

CONTACTS AND LOCATIONS:
Overall Officials: Bruno LABEILLE, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France